CLINICAL TRIAL: NCT07360873
Title: Effect of Eccentric Exercises of Calf Muscles Versus Heel Insole Lift on Pain, Range of Motion, and Function in Football Players With Achilles Tendinopathy
Brief Title: Eccentric Exercises Versus Heel Insole Lift for Achilles Tendinopathy in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adnan Hashim (Other)
Collaborators: University of Lahore Hospital (ULH) (Network)
Responsible Party: Sponsor-Investigator, Adnan Hashim, Doctor of Physical Therapy Student, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRI/IREB/26/01/0035
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Achilles Tendinopathy (AT)
Keywords: Achilles Tendinopathy; Eccentric Exercise; Heel Lift; Calf Muscle; Football Players; Sports Rehabilitation; Physiotherapy; Ankle Function

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups to receive either an eccentric calf muscle exercise program or heel insole lifts for a 12-week intervention period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation to minimize assessment bias. Participants and care providers were not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric Calf Muscle Exercise Group (Experimental): Participants assigned to this arm received a structured eccentric calf muscle exercise program based on Alfredson's protocol for the management of Achilles tendinopathy.
  Interventions: Other: Eccentric Calf Muscle Exercises
- Heel Insole Lift Group (Active Comparator): Participants assigned to this arm were provided with heel insole lifts and instructed to use them during daily activities throughout the intervention period.
  Interventions: Device: Heel Insole Lift

INTERVENTIONS:
Other: Eccentric Calf Muscle Exercises — Eccentric calf muscle exercises were performed according to Alfredson's protocol. Participants completed three sets of fifteen repetitions, twice daily, seven days per week for 12 weeks. Exercises were performed on a step with the knee extended and flexed to target the gastrocnemius and soleus muscles. Resistance was progressively increased as pain decreased.
  Arms: Eccentric Calf Muscle Exercise Group
Device: Heel Insole Lift — Participants were provided with prefabricated heel insole lifts (approximately 12 mm) based on shoe size and instructed to wear them continuously in their regular footwear during daily activities for a 12-week period.
  Arms: Heel Insole Lift Group

SUMMARY:
Achilles tendinopathy is a common overuse injury in football players and is associated with pain, stiffness, and reduced functional performance. Conservative treatment options such as eccentric calf muscle exercises and heel insole lifts are frequently used in rehabilitation; however, evidence comparing their effectiveness remains limited.

This randomized controlled trial compared the effects of eccentric calf muscle exercises and heel insole lifts on pain, ankle range of motion, and functional outcomes in male football players with Achilles tendinopathy. Participants were randomly assigned to one of two intervention groups. One group performed a structured eccentric calf muscle exercise program, while the other group used heel insole lifts during daily activities.

Outcomes related to pain intensity, functional ability, calf muscle performance, and ankle range of motion were assessed at baseline and after completion of a 12-week intervention period. The results of this study aim to support evidence-based rehabilitation strategies for the management of Achilles tendinopathy in football players.

DETAILED DESCRIPTION:
This study was a single-blinded, randomized controlled trial conducted after obtaining ethical approval from the institutional ethics review committee. Male football players aged 18 to 30 years with clinically diagnosed Achilles tendinopathy were recruited from football clubs in Lahore, Pakistan, using a non-probability convenience sampling technique. Participants who met the eligibility criteria were randomly allocated into two parallel intervention groups using a lottery method.

Participants in the experimental group received an eccentric calf muscle exercise program based on Alfredson's protocol. The exercises were performed on a step with the knee extended and slightly flexed to target the gastrocnemius and soleus muscles, respectively. The protocol consisted of three sets of fifteen repetitions, performed twice daily, seven days per week, over a 12-week period. Body weight was used as resistance, and additional external load was progressively added as pain decreased.

Participants in the control group were provided with prefabricated heel insole lifts and instructed to wear them continuously in their regular footwear during daily activities throughout the 12-week intervention period.

Outcome measures were assessed at baseline and after completion of the intervention period. These included pain intensity, functional ability, calf muscle endurance, and ankle dorsiflexion range of motion. The study was conducted in accordance with ethical principles, and written informed consent was obtained from all participants prior to enrollment. The findings of this study are intended to contribute to evidence-based sports rehabilitation practices for the management of Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male football players aged 18 to 30 years
* Clinical diagnosis of Achilles tendinopathy
* Achilles tendon pain for at least one month
* Pain intensity of 3 or higher on the Visual Analogue Scale
* Pain aggravated by weight-bearing activities
* Able to understand English and complete questionnaires
* Willing to avoid other treatments for Achilles tendinopathy during the 12-week study period

Exclusion Criteria:

* Lower limb injury within the past 6 months
* Previous Achilles tendon rupture or surgery
* Chronic ankle instability
* Recent use of eccentric exercises or heel insole lifts
* Metabolic or endocrine disorders
* Current use of medications other than paracetamol
* Unwillingness to comply with the study protocol

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Functional Ability (Victorian Institute of Sports Assessment-Achilles, VISA-A) | Baseline and at 12 weeks
  Functional status was assessed using the Victorian Institute of Sports Assessment-Achilles (VISA-A) questionnaire. Scores range from 0 to 100, with higher scores indicating better function (less severe symptoms).
Pain Intensity (Visual Analogue Scale, VAS) | Baseline and at 12 weeks
  Pain intensity was assessed using the Visual Analogue Scale (VAS), a 100-mm scale ranging from 0 (no pain) to 100 (worst imaginable pain). Higher scores indicate worse pain. Outcome is reported in millimeters (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Hashim, DPT, Principal Investigator — Department of Physical Therapy, The University of Lahore
Locations (1):
- FAME Football Club, Model Town, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study was conducted as an academic research project. The informed consent obtained from participants did not include provisions for public data sharing, and the dataset contains sensitive personal health information. Data will be stored securely and used only for academic and research purposes in accordance with institutional ethics approval.

REFERENCES:
- [Background] Zhang BM, Zhong LW, Xu SW, Jiang HR, Shen J. Acupuncture for chronic Achilles tendnopathy: a randomized controlled study. Chin J Integr Med. 2013 Dec;19(12):900-4. doi: 10.1007/s11655-012-1218-4. Epub 2012 Dec 21. PMID 23263998
- [Background] van der Vlist AC, Winters M, Weir A, Ardern CL, Welton NJ, Caldwell DM, Verhaar JAN, de Vos RJ. Which treatment is most effective for patients with Achilles tendinopathy? A living systematic review with network meta-analysis of 29 randomised controlled trials. Br J Sports Med. 2021 Mar;55(5):249-256. doi: 10.1136/bjsports-2019-101872. Epub 2020 Jun 10. PMID 32522732
- [Background] Stevens M, Tan CW. Effectiveness of the Alfredson protocol compared with a lower repetition-volume protocol for midportion Achilles tendinopathy: a randomized controlled trial. J Orthop Sports Phys Ther. 2014 Feb;44(2):59-67. doi: 10.2519/jospt.2014.4720. Epub 2013 Nov 21. PMID 24261927
- [Background] Stasinopoulos D, Manias P. Comparing two eccentric exercise programmes for the management of Achilles tendinopathy. A pilot trial. J Bodyw Mov Ther. 2013 Jul;17(3):309-15. doi: 10.1016/j.jbmt.2012.11.003. Epub 2012 Dec 12. PMID 23768274
- [Background] Siu WL, Chan CH, Lam CH, Lee CM, Ying M. Sonographic evaluation of the effect of long-term exercise on Achilles tendon stiffness using shear wave elastography. J Sci Med Sport. 2016 Nov;19(11):883-887. doi: 10.1016/j.jsams.2016.02.013. Epub 2016 Mar 11. PMID 26996945
- [Background] Silbernagel KG, Hanlon S, Sprague A. Current Clinical Concepts: Conservative Management of Achilles Tendinopathy. J Athl Train. 2020 May;55(5):438-447. doi: 10.4085/1062-6050-356-19. Epub 2020 Apr 8. PMID 32267723
- [Background] Silbernagel KG, Crossley KM. A Proposed Return-to-Sport Program for Patients With Midportion Achilles Tendinopathy: Rationale and Implementation. J Orthop Sports Phys Ther. 2015 Nov;45(11):876-86. doi: 10.2519/jospt.2015.5885. Epub 2015 Sep 21. PMID 26390272
- [Background] Shih, K.-S., Chen, P.-Y., Yeh, W.-L., Ma, H.-L., Farn, C.-J., Hou, C.-H., Peng, W.-C., & Wang, H.-K. (2021). Modified Ankle Joint Neuromechanics during One-Legged Heel Raise Test after an Achilles Rupture and Its Associations with Jumping. Applied Sciences, 11(5), 2227.
- [Background] Radovanovic G, Bohm S, Peper KK, Arampatzis A, Legerlotz K. Evidence-Based High-Loading Tendon Exercise for 12 Weeks Leads to Increased Tendon Stiffness and Cross-Sectional Area in Achilles Tendinopathy: A Controlled Clinical Trial. Sports Med Open. 2022 Dec 20;8(1):149. doi: 10.1186/s40798-022-00545-5. PMID 36538166
- [Background] Rabusin CL, Menz HB, McClelland JA, Evans AM, Malliaras P, Docking SI, Landorf KB, Gerrard JM, Munteanu SE. Efficacy of heel lifts versus calf muscle eccentric exercise for mid-portion Achilles tendinopathy (HEALTHY): a randomised trial. Br J Sports Med. 2021 May;55(9):486-492. doi: 10.1136/bjsports-2019-101776. Epub 2020 Sep 28. PMID 32988930
- [Background] Rabusin CL, Menz HB, McClelland JA, Evans AM, Landorf KB, Malliaras P, Docking SI, Munteanu SE. Efficacy of heel lifts versus calf muscle eccentric exercise for mid-portion Achilles tendinopathy (the HEALTHY trial): study protocol for a randomised trial. J Foot Ankle Res. 2019 Mar 21;12:20. doi: 10.1186/s13047-019-0325-2. eCollection 2019. PMID 30949243
- [Background] Prudencio DA, Maffulli N, Migliorini F, Serafim TT, Nunes LF, Sanada LS, Okubo R. Eccentric exercise is more effective than other exercises in the treatment of mid-portion Achilles tendinopathy: systematic review and meta-analysis. BMC Sports Sci Med Rehabil. 2023 Jan 26;15(1):9. doi: 10.1186/s13102-023-00618-2. PMID 36698184
- [Background] O'Neill S, Watson PJ, Barry S. WHY ARE ECCENTRIC EXERCISES EFFECTIVE FOR ACHILLES TENDINOPATHY? Int J Sports Phys Ther. 2015 Aug;10(4):552-62. PMID 26347394
- [Background] Martin RL, Chimenti R, Cuddeford T, Houck J, Matheson JW, McDonough CM, Paulseth S, Wukich DK, Carcia CR. Achilles Pain, Stiffness, and Muscle Power Deficits: Midportion Achilles Tendinopathy Revision 2018. J Orthop Sports Phys Ther. 2018 May;48(5):A1-A38. doi: 10.2519/jospt.2018.0302. PMID 29712543
- [Background] Maffulli N, Longo UG, Kadakia A, Spiezia F. Achilles tendinopathy. Foot Ankle Surg. 2020 Apr;26(3):240-249. doi: 10.1016/j.fas.2019.03.009. Epub 2019 Apr 18. PMID 31031150
- [Background] Leung WKC, Chu KL, Lai C. Sonographic evaluation of the immediate effects of eccentric heel drop exercise on Achilles tendon and gastrocnemius muscle stiffness using shear wave elastography. PeerJ. 2017 Jul 19;5:e3592. doi: 10.7717/peerj.3592. eCollection 2017. PMID 28740756
- [Background] Lee KKW, Ling SKK, Yung PSH. Controlled trial to compare the Achilles tendon load during running in flatfeet participants using a customized arch support orthoses vs an orthotic heel lift. BMC Musculoskelet Disord. 2019 Nov 13;20(1):535. doi: 10.1186/s12891-019-2898-0. PMID 31722697
- [Background] Karamat MS, Jamil A. Comparative effects of myofascial release with and without eccentric resistance on pain, range of motion, and functional disability in patients with Achilles tendinopathy. J Bodyw Mov Ther. 2024 Oct;40:1066-1071. doi: 10.1016/j.jbmt.2024.07.029. Epub 2024 Jul 9. PMID 39593413
- [Background] Habets B, van Cingel RE. Eccentric exercise training in chronic mid-portion Achilles tendinopathy: a systematic review on different protocols. Scand J Med Sci Sports. 2015 Feb;25(1):3-15. doi: 10.1111/sms.12208. Epub 2014 Mar 20. PMID 24650048
- [Background] Griffin, C. (2023). Achilles tendon injury rehabilitation and lower limb biomechanics Université Côte d'Azur].
- [Background] Gerdesmeyer L, Mittermayr R, Fuerst M, Al Muderis M, Thiele R, Saxena A, Gollwitzer H. Current evidence of extracorporeal shock wave therapy in chronic Achilles tendinopathy. Int J Surg. 2015 Dec;24(Pt B):154-9. doi: 10.1016/j.ijsu.2015.07.718. Epub 2015 Aug 29. PMID 26327530
- [Background] Engh, L., Fall, M., Hennig, M., & Söderlund, A. (2003). Intra-and inter-rater reliability of goniometric method of measuring head posture. Physiotherapy Theory and Practice, 19(3), 175-182.
- [Background] de Jonge S, van den Berg C, de Vos RJ, van der Heide HJ, Weir A, Verhaar JA, Bierma-Zeinstra SM, Tol JL. Incidence of midportion Achilles tendinopathy in the general population. Br J Sports Med. 2011 Oct;45(13):1026-8. doi: 10.1136/bjsports-2011-090342. PMID 21926076
- [Background] Cuyul-Vasquez I, Alvarez E, Riquelme A, Zimmermann R, Araya-Quintanilla F. Effectiveness of Unilateral Training of the Uninjured Limb on Muscle Strength and Knee Function of Patients With Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-Analysis of Cross-Education. J Sport Rehabil. 2022 Mar 12;31(5):605-616. doi: 10.1123/jsr.2021-0204. Print 2022 Jul 1. PMID 35279020
- [Background] Couppe C, Svensson RB, Silbernagel KG, Langberg H, Magnusson SP. Eccentric or Concentric Exercises for the Treatment of Tendinopathies? J Orthop Sports Phys Ther. 2015 Nov;45(11):853-63. doi: 10.2519/jospt.2015.5910. Epub 2015 Oct 15. PMID 26471850
- [Background] Chukwuemeka, U., Anyoku, C., Onwuakagba, I., & Akobundu, U. (2022). Prevalence and Risk Factors of Achilles Tendinopathy among University Soccer Players. Int J Sports Exerc Med, 8, 223.
- [Background] Bourke J, Munteanu S, Garofolini A, Taylor S, Malliaras P. Efficacy of heel lifts for mid-portion Achilles tendinopathy (the LIFT trial): study protocol for a randomised controlled trial. Trials. 2024 May 24;25(1):345. doi: 10.1186/s13063-024-08185-8. PMID 38790025
- [Background] Beyer R, Kongsgaard M, Hougs Kjaer B, Ohlenschlaeger T, Kjaer M, Magnusson SP. Heavy Slow Resistance Versus Eccentric Training as Treatment for Achilles Tendinopathy: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1704-11. doi: 10.1177/0363546515584760. Epub 2015 May 27. PMID 26018970
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Aiyegbusi, A., Owoeye, I., Balogun, O., Fapojuwo, O., & Akinloye, O. (2021). Prevalence of Achilles Tendinopathy and Associated Selected Intrinsic Risk Factors among Nigerian Footballers. Muscles, Ligaments & Tendons Journal (MLTJ), 11(1).